CLINICAL TRIAL: NCT06054659
Title: A Randomized Controlled Open-label Study Comparing the Use of Real-time Continuous Glucose Monitoring (Rt-CGM) to Point of Care Testing (POCT) for Glycemic Monitoring in Patients Post-hospitalization for Diabetic Foot Ulcers.
Brief Title: CGM and DFU Healing Post-discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maya Fayfman, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006202; R03DK137007-01 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot; Diabetes Type 2 With Diabetic Ulcer of Toe, Skin Breakdown
Keywords: Continuous Glucose Monitoring (CGM) system; Time in Range; Fingerstick blood glucose testing; Wound healing; Real time - Continuous glucose monitoring
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Real time - Continuous glucose monitoring (Experimental): Participants will wear a CGM sensor in the abdomen or arm, placed by a study team before hospital discharge. Participants will have instructions on how to monitor BG with the CGM device and will use their glucometer and do fingersticks as needed for CGM calibration.
  Interventions: Device: Real Time Continuous Glucose Monitoring (rt-CGM); Other: Fingerstick blood glucose (FBG) monitoring; Behavioral: Diabetes Education
- Fingerstick blood glucose (FBG) monitoring (Active Comparator): Participants randomized to this group will monitor blood glucose by performing fingersticks, they will also have the application of CGM but will not be given the receiver to allow for self-monitoring. CGM will only be applied by the research team for monitoring over a 14-day interval at baseline, week 4, week 8, and week 12. Blinding will continue throughout the study. This group will receive training only in home BG monitoring with FBG.
  Interventions: Other: Fingerstick blood glucose (FBG) monitoring; Behavioral: Diabetes Education

INTERVENTIONS:
Device: Real Time Continuous Glucose Monitoring (rt-CGM) — Participants randomized to rt-CGM will have CGM placed before hospital discharge. They will also receive teaching from the research team on the proper use of their CGM sensor and reader. The study team will provide CGM devices, but subjects may use their glucometer for FBG testing as needed for CGM calibration.
  Other Names: Intervention Group
  Arms: Real time - Continuous glucose monitoring
Other: Fingerstick blood glucose (FBG) monitoring — Participants will use their own glucometer for FBG testing as advised by their treating provider (usually primary care or diabetes doctor).
  Other Names: Standard of Care (SOC) capillary glucose test
Behavioral: Diabetes Education — Participants will receive standard-of-care diabetes education with a certified diabetes educator (CDE) prior to discharge (with the approval of the treating inpatient team).

SUMMARY:
The purpose of this study is to look at the benefits of using a Continuous Glucose Monitoring (CGM) system compared with standard-of-care testing for patients with type 2 diabetes and diabetic foot ulcers (DFU) and how this will improve wound healing.

The CGM system allows medical staff and patients with diabetes to monitor and make treatment decisions to improve glucose control, without the need for performing fingersticks. Hence, the use of CGM will decrease the painful and burdensome task of performing finger sticks several times per day and may prevent low blood glucose in patients with diabetes.

DETAILED DESCRIPTION:
The goals of this study are to compare differences in patients with diabetic foot ulcer (DFU) wound healing using continuous glucose monitor (CGM) and point of care testing (POCT) at 16 weeks post-hospital discharge. The study is important to support the limited data available to optimize glycemic control DFU healing and the use of CGM. Patients with type 2 diabetes (T2D) and HbA1c > 8.5% admitted to general medicine and surgery services with diabetic foot ulcers will be approached for study participation.

After completing the informed consent process, patients will be randomized 1:1 to glucose monitoring with real-time CGM (rt-CGM) or POCT. Before discharge, participants in the rt-CGM group will have CGM applied by the research team with instructions on how to monitor blood glucose (BG) with the CGM device. Participants enrolled in the POCT group will have the application of a blinded CGM that will monitor glycemic control, but results will not be visible to the participant, clinical team, or research providers. Participants will receive standard diabetes education. Participants will be scheduled for research visits at 4, 8, 12, and 16 weeks. CGM sensors will be provided at these visits with a review of application, monitoring, and removal. Subjects in both groups will not receive specific guidelines on medication or other interventions. At the end of the 16-week study period, an assessment of final wound outcomes will be made by either the podiatry or infectious diseases collaborators (one of whom will have already been following the patient clinically) during one of the routine clinical visits. Photos of the ulcer site will be taken at the 16-week study visit, and the outcome will be reported by the treating wound care provider and adjudicated by a member of the study team who is blinded to the patient's clinical information and intervention arm. Participants will complete surveys to assess patient-reported outcomes relating to depression, CGM satisfaction, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over with type 2 diabetes admitted to the hospital with diabetic foot ulceration with or without infection (cellulitis or osteomyelitis)
* HbA1c >= 8.0% at the time of enrollment
* Treatment of diabetic foot ulcer with medical management and/or a single toe amputation
* Patients with prior amputation at or below the ankle may be enrolled if they develop an ulceration in the foot that is not felt to be a surgical wound from prior amputation, defined as a healed surgical site for at least 6 weeks after the surgery before the onset of the new ulceration
* Wound, Ischemia, foot Infection (WIfI) score of 1-3
* Duration of DFU less than 1 year
* Able and willing to use continuous glucose monitoring technology independently or with the assistance of a close relative or caretaker

Exclusion Criteria:

* Age < 18 years
* Homelessness or anticipated to have unstable housing after discharge
* A WIfI score of 4, denoting a very high risk for major amputation (above or below the knee) and very low odds of healing within 12 months
* Any amputation more extensive than just a single toe during index hospitalization
* Patients with type 1 diabetes
* Participants enrolled in another interventional clinical trial (including during the run-in period).
* Inability to participate in the informed consent process for any reason
* Female subjects who are pregnant or breastfeeding at the time of enrollment in the study
* Subjects planning to use CGM technology independent of the study following discharge
* Subjects unwilling to wear a CGM device and/or monitor blood glucose with FBG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
DFU wound healing rates | up to 16 weeks post-discharge
  Number of participants with DFU wound healing rates in both groups
Time to DFU healing | up to 16 weeks post-discharge
  DFU healing will be assessed by two investigators blinded to the study intervention

SECONDARY OUTCOMES:
Change in patient reported World Health Organization Well-Being Index | Baseline and 16 weeks post-discharge
  The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, with 0 representing the worst possible and 25 representing the best possible quality of life. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents the worst possible, whereas a score of 100 represents the best possible quality of life. A score below 13 indicates poor well-being and is an indication for testing for depression. In order to monitor possible changes in wellbeing, the percentage score is used. A 10% difference indicates a significant change.
Change in patient reported diabetes distress scores (DDS) | Baseline and 16 weeks post-discharge
  The DDS yields a total diabetes distress score plus 4 subscale scores, each addressing a different kind of distress. To score, simply sum the patient's responses to the appropriate items and divide by the number of items in that scale. Current research suggests that a mean item score of 2.0 - 2.9 should be considered 'moderate distress,' and a mean item score > 3.0 should be considered 'high distress.' Current research also indicates that associations between DDS scores and behavioral management and biological variables (e.g., A1C) occur with DDS scores of > 2.0. Clinicians may consider moderate or high distress worthy of clinical attention, depending on the clinical context.
Change in patient reported CGM satisfaction (CGM-SAT) | Baseline and 16 weeks post-discharge
  CGM-SAT: This 44-item questionnaire was designed to measure the impact of using CGM on diabetes management and family relationships and on satisfaction with the emotional, behavioral, and cognitive effects of CGM use. Participants rate their agreement or disagreement on a 5-point Likert scale (1 = strongly agree; 5 = strongly disagree) with each of 44 potential positive or negative effects of the use of the rated CGM device. Higher scores reflect a more favorable impact of, and satisfaction with, CGM use.
Change in patient reported Glucose Monitoring Survey (GMS) | Baseline and 16 weeks post-discharge
  GMS is a 22-item scale constructed for this trial that quantifies respondents' satisfaction with and therapeutic impact of the glucose monitoring systems that they were currently using (SMBG alone or with CGM). The 22 two-part items ask the respondent to evaluate "Is this a problem now?" and then "How has it changed in the past 6 months?" Response options for the "Problem" questions range from 1 = "a lot" to 4 = "not at all," while those for the "Change" questions range from 1 = "worse" to 3 = "better." Higher scores on the "Problem" questions indicate more positive views of the rated glucose monitoring system. Higher scores on the "Change" questions indicate greater perceived improvement.
Frequency of medication adjustments | Up to 16 weeks post discharge
  The frequency of medication adjustments including initiation of new non-insulin-based therapy, basal and/or prandial insulin therapy, and/or dose adjustments will be documented during study participation.
Glycemic variability | Baseline and 16 weeks post-discharge
  Glycemic variability (GV) will be assessed by coefficient of variation (CV) and standard deviation from baseline and 12 weeks. Based on the published literature, the 2017 international consensus statement on the use of CGM suggested that 'stable glucose levels are defined as a CV <36% and unstable glucose levels are defined as CV ≥36%
Relationship of time in range (TIR) and likelihood of healing | Up to 16 weeks post discharge
  Time in Range (%TIR) is the percentage of time that a person spends with their blood glucose levels in a target range (70-180 mg/dL). A time-to-event (TTE) analysis will be conducted with the primary outcome based on time in range (%TIR) stratification among all study subjects. The stratification will be done for groups where %TIR ≥ 50 and %TIR < 50%.
Relationship of time below range (%TBR) and likelihood of healing | Up to 16 weeks post discharge
  Healing rate compared to each %TBR level 1 (54 - < 70 mg/dL); %TBR Level 2 (BG<54 mg/dL)
Relationship of time above range (%TAR) and likelihood of healing | Up to 16 weeks post discharge
  Healing rate compared to each %TAR level 1 (BG >180 - 250 mg/dL); %TAR level 2 (BG >250 mg/dL)
Relationship of glycemic variability and the likelihood of healing | Up to 16 weeks post discharge
  Healing rate compared to GV

CONTACTS AND LOCATIONS:
Overall Officials: Maya Fayfman, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available for sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Individual participant data will be made available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Individual participant data will be made available for sharing with researchers who provide a methodologically sound proposal. The proposal should be directed to maya.fayfman@emory.edu. To gain access, data requestors will need to sign a data access agreement.